CLINICAL TRIAL: NCT06747611
Title: Evaluation of Microbiota Transplant Therapy in Patients With Alopecia Areata
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DERM-2022-30819
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — Vancomycin; Neomycin; monooxyethylene trimethylolpropane tristearate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alopecia Areata study group (Experimental): randomized to receive antibiotics and MTT oral capsule
  Interventions: Drug: Vancomycin, Neomycin and MTT capsules
- Alopecia Areata control group (Placebo Comparator): randomized to receive placebo antibiotics and placebo MTT oral capsule
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Vancomycin, Neomycin and MTT capsules — patients will take 2 capsules per day for 14 days. These patients will then be clinically followed for a period of 24 weeks.
  Arms: Alopecia Areata study group
Drug: Placebo capsules — patients will take 2 capsules per day for 14 days. These patients will then be clinically followed for a period of 24 weeks.
  Arms: Alopecia Areata control group

SUMMARY:
Alopecia Areata (AA) is among the most highly prevalent human autoimmune diseases, leading to disfiguring hair loss due to the collapse of immune privilege of the hair follicle and subsequent autoimmune attack. AA affects about 5.3 million people in the United States alone, including males and females across all ethnic groups, with a lifetime risk of 2.1%. Autoimmunity develops against the hair follicle, resulting in non-scarring hair loss that may begin as patches that can coalesce and progress to cover the entire scalp (alopecia totalis) or eventually the entire body (alopecia universalis). In AA, there is no permanent destruction of the hair follicle, and regrowth remains possible. Treatment options for AA include intralesional steroids, topical anthralin, allergic contact dermatitis with diphencyprone (DPCP), dinitrochlorobenzene (DNCB), or squaric acid dibutyl ester (SADBE), and recently janus kinase ( JAK) inhibitors. Despite the recent approval of JAKs for the treatment of extensive alopecia areata, some patients are treatment resistant, suffer relapses, or cannot take an oral immunosuppressive medication.

This study will attempt to elucidate the pre-treatment and post treatment skin and gut microbiome composition to determine whether specific bacterial species may correlate with disease or treatment response. To determine the effects of MTT on immune cell composition and activation systemically and locally in the skin, we will analyze major immune cell populations in peripheral blood samples and collect skin biopsies for histopathology and next generation sequencing analyses. Further, to determine if changes in immune cell populations affect the inflammatory response, we will profile inflammatory cytokines. To identify if changes in the gut microbiota influence the metabolic signature in AA, we will also perform untargeted metabolomics in stool gut microbiome samples and in plasma. Altogether, this comprehensive approach aims to identify the pathogenic immunological mechanisms associated with microbiome composition correlated to pre-treatment disease, post-treatment response, and any non-responders to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 75 years of age with moderate to severe alopecia areata (SALT score >30%).
* Patients with a diagnosis of patch type alopecia areata, totalis, or universalis..
* Duration of hair loss >=3 months..
* No evidence of active, ongoing regrowth present at baseline.
* Females of childbearing potential must have a negative urine or serum pregnancy test at screening and immediately prior to MTT.
* Females of childbearing potential must agree to use an effective form of contraception from 14 days prior to study antibiotics through at least 30 days after MTT. Acceptable forms of contraception include oral or intramuscular contraceptives, intrauterine devices, surgical sterilization.
* Participants are not enrolled in another clinical study.
* If undergoing treatment with a JAK inhibitor, participant is willing to discontinue treatment for 1 month prior to enrollment and throughout the duration of the study.

Exclusion Criteria:

* Active gastrointestinal infection at time of enrollment.
* Having been administered antibiotics in the last 48 hours.
* Patients will be eligible to enroll if antibiotic therapy is discontinued for at minimum 48 hours prior to treatment..
* Requires continued antibiotic use
* Allergy to study antibiotics (vancomycin, neomycin).
* Known or suspected severe gastrointestinal dysmotility disorder, e.g., gastroparesis, pseudo-obstruction, scleroderma with gastrointestinal involvement
* Ileus or small bowel obstruction.
* Major gastrointestinal surgery (e.g., significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy.
* History of total colectomy.
* Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy.
* Unable or unwilling to comply with protocol requirements.
* Expected life expectancy < 6 months.
* Previous MTT or microbiome-based products at any time excluding this study.
* History of severe anaphylactic or anaphylactoid food allergy.
* Solid organ transplant recipients 90 days post-transplant or on active treatment for rejection.
* A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study.
* History of or existing skin diseases affecting the scalp such as psoriasis or seborrheic dermatitis and patients with evidence of infection or skin cancer in the treated areas.
* Patients in whom the diagnosis of alopecia areata is questionable.
* Patients in whom regrowth is present/evident at baseline in the areas to be treated.
* Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma of the skin) which in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections.
* Patients unwilling or unable to discontinue treatments known to affect hair regrowth in alopecia areata.
* Patients who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, DPCP (diphenylcycloprophenone), protopic, minoxidil, JAK inhibitors or other medication which in the opinion of the investigator may affect hair regrowth, within one month of the baseline visit..
* Patients determined by the investigator to have extreme diets..
* Pregnant and breastfeeding females..

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Engraftment | Week 8
  Proportion of patients achieving donor microbiota engraftment measured at 8 weeks post treatment.

SECONDARY OUTCOMES:
Hair regrowth | 8, 16, 24, 26, 34, 42, 50 and 54 weeks post treatment
  Percent hair regrowth from baseline determined by SALT measurements following 8, 16, 24, 26, 34, 42, 50 and 54 weeks post treatment.
efficacy measure 2 | 6 months post therapy
  Timing of relapse in responders followed for 6 months post therapy.
SALT Score | Week 24
  Proportion of patients in the treatment versus placebo group achieving SALT score of <50% at week 24
safety outcome 2 | day 30
  Proportion of participants with a SAE through day 30 (±3 days) after MTT.
safety outcome 3 | day 30
  Proportion of participants with newly acquired transmissible infectious diseases which are considered adverse events of special interest (AESI) through day 30 (±3 days) after MTT.
safety outcome 1 | day 30
  Proportion of participants with an AE through day 30 (±3 days) after MTT.
Week 4 AEs | Week 4
  Proportion of participants with an AE through week 4 (±5 days) after MTT.
Week 4 SAEs | Week 4
  Proportion of participants with an SAE through week 4 (±5 days) after MTT.
Month 6 SAEs | Month 6
  Proportion of participants with a SAE at month 6 (±14 days) after randomization.
Month 12 SAEs | Month 12
  Proportion of participants with a SAE at month 12 (±14 days) after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States